CLINICAL TRIAL: NCT07006922
Title: Can a Platelet-Rich Plasma Covering Layer Reduce Urethrocutaneous Fistula Rate After Distal Penile Hypospadias Repair Using the STAR Technique: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelghany, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS*225-2024
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2024-07

CONDITIONS: Hypospadias; Pediatric Urology
Keywords: Platelet-Rich Plasma; Hypospadias Repair; Urethrocutaneous Fistula; Pediatric Urology.; STAR Technique
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STAR+ PRP (Experimental): underwent repair using the STAR technique with an additional PRP layer over the neourethra
  Interventions: Procedure: hypospadias repair using the STAR technique with PRP as protective layer
- STAR only (Experimental): received the STAR repair without PRP
  Interventions: Procedure: hypospadias repair using the STAR technique

INTERVENTIONS:
Procedure: hypospadias repair using the STAR technique with PRP as protective layer — the STAR technique involves anatomical reassembly of penile tissues guided by the topography of the glans and corpus spongiosum (the exclusive zipping-up of the unfolded spongiosal plate). A fine-tipped tenotomy scissor used for dissection, starting at the apex of the hypoplastic "V" and extending into the ventral edges of the hooded prepuce on each side, following the demarcation lines. Then, a midline cutting back of the ventral hypoplastic urothelial sheet from the hypospadias meatus to the point of spongiosal bifurcation was made . Excision of the hypoplastic skin ridge all the way from the point of bifurcation till each ipsilateral ventral endpoint of the glanular meatal marks to maximize the epithelialized endoluminal surface of the newly zipped-up spongiosal plate. An interrupted single -layedred spongioplasty ( zipper closure) using 6/0 Vicryl Absorbable sutures (13mm needle, Ethicon Inc, Somerville, New Jersey) is applied over a naeleton catheter . Lastly, the glansplasty is d
  Arms: STAR+ PRP
Procedure: hypospadias repair using the STAR technique — the STAR technique involves anatomical reassembly of penile tissues guided by the topography of the glans and corpus spongiosum (the exclusive zipping-up of the unfolded spongiosal plate). A fine-tipped tenotomy scissor used for dissection, starting at the apex of the hypoplastic "V" and extending into the ventral edges of the hooded prepuce on each side, following the demarcation lines. Then, a midline cutting back of the ventral hypoplastic urothelial sheet from the hypospadias meatus to the point of spongiosal bifurcation was made . Excision of the hypoplastic skin ridge all the way from the point of bifurcation till each ipsilateral ventral endpoint of the glanular meatal marks to maximize the epithelialized endoluminal surface of the newly zipped-up spongiosal plate. An interrupted single -layedred spongioplasty ( zipper closure) using 6/0 Vicryl Absorbable sutures (13mm needle, Ethicon Inc, Somerville, New Jersey) is applied over a naeleton catheter . Lastly, the glansplasty is d
  Arms: STAR only

SUMMARY:
Methods We conducted a prospective randomized controlled study at the Pediatric Urology Department of Cairo University Specialized Pediatric Hospital between July 2024 and January 2025 . The study included boys undergoing primary repair of distal penile hypospadias. Ethical approval was obtained from the institution's review board, and informed consent was secured from the parents or legal guardians of all participants.

The study included distal penile hypospadias (glandular, coronal, or subcoronal meatus). Exclusion criteria were: proximal or mid-penile hypospadias, any history of prior hypospadias repair, bleeding or coagulation disorders and other significant genitourinary anomalies.

The participants were randomly allocated into two equal groups using simple randomization (sealed envelope method). Group A (PRP group) underwent repair with the STAR technique plus an intermediate PRP covering layer. Group B (Control group) underwent repair using the same technique but without PRP. All surgeries were performed by the same pediatric urologist, an experienced surgeon in hypospadias repair, to eliminate inter-surgeon variability.

All patients were operated on under general anesthesia with caudal block analgesia. A standard STAR hypospadias repair was carried out in each case as described by Seleim (10). In brief, the STAR technique involves anatomical reassembly of penile tissues guided by the topography of the glans and corpus spongiosum (the exclusive zipping-up of the unfolded spongiosal plate). A fine-tipped tenotomy scissor used for dissection, starting at the apex of the hypoplastic "V" and extending into the ventral edges of the hooded prepuce on each side, following the demarcation lines. Then, a midline cutting back of the ventral hypoplastic urothelial sheet from the hypospadias meatus to the point of spongiosal bifurcation was made . Excision of the hypoplastic skin ridge all the way from the point of bifurcation till each ipsilateral ventral endpoint of the glanular meatal marks to maximize the epithelialized endoluminal surface of the newly zipped-up spongiosal plate. An interrupted single -layedred spongioplasty ( zipper closure) using 6/0 Vicryl Absorbable sutures (13mm needle, Ethicon Inc, Somerville, New Jersey) is applied over a naeleton catheter . Lastly, the glansplasty is done using 3 slanting sutures. In Group A, before skin closure, a PRP layer was applied over the neourethra, whereas in Group B the repair proceeded directly to skin closure without PRP.

PRP Preparation and Application In Group A patients, approximately 5-10 mL of the child's blood was drawn from a peripheral vein at the start of the operation. The blood was collected into a sterile tube without anticoagulant additives and immediately centrifuged at ~3000 rpm for 20 minutes. This process separated the blood into three components: an upper platelet-poor plasma, a middle platelet-rich plasma, and a bottom red blood cell layer. The platelet-rich plasma fraction was then isolated. After the neourethra was constructed and prior to skin closure, the PRP was applied directly as a liquid/gel onto the repair site covering the neourethra. In a few minutes, PRP forms a clot-like gel layer. No additional dartos or fascia flaps were used in either group, in keeping with the STAR technique's usual practice.

Postoperative Care and Follow-up All patients had a compressive dressing applied, which was removed on the third postoperative day. A urethral stent catheter was left in place to divert urine; this was kept for 7 days postoperatively. Broad-spectrum prophylactic antibiotics were given while the catheter was in situ. Parents were instructed on catheter care and advised to ensure the child avoided straddling activities.

After catheter removal, the urinary stream was observed to ensure it was not deviated or weak. Patients were followed up weekly for at least 4 weeks after surgery, and then monthly up to 3 months. At each follow-up visit, the penis was examined for any complications including urethrocutaneous fistula, meatal stenosis, wound infection, glans dehiscence, and persistent edema or flap necrosis.

Cosmetic and functional outcomes were evaluated at the 1-month visit and again at 3 months using the HOSE score, which assigns points for meatal location, meatal shape, urinary stream, erection straightness, and overall appearance. A higher HOSE score (maximum 16) indicates a more favorable outcome.

Outcome Measures The primary outcome measure was the occurrence of urethrocutaneous fistula within the follow-up period. Key secondary outcomes included incidence of other complications (edema, infection, meatal stenosis, glans dehiscence), the operative time (skin-to-skin surgical duration in minutes), and the cosmetic outcome (HOSE score and meatal configuration).

Statistical Analysis Data were analyzed using the statistics software, SPSS software (IBM SPSS, v25). Continuous variables like age and operative time were not normall

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with distal penile hypospadias, primary or fresh cases will be selected and circumcised or uncircumcised are included

Exclusion Criteria:

* Pediatric patients with other types of hypospadias, distal penile hypospadias who has history of previous surgical trail

Ages: 6 Months to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
urethrocutaneous fistula | 4 weeks

SECONDARY OUTCOMES:
postoperative complications (edema, infection, meatal stenosis), operative time, and cosmetic outcome using the Hypospadias Objective Scoring Evaluation (HOSE). | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt